CLINICAL TRIAL: NCT04531150
Title: A Single Center, Phase I, Double-Blind, Placebo-Controlled Evaluation of the Safety, Tolerability, and Pharmacokinetics of Single Ascending Oral Doses of INV-101 in Healthy Male and Female Subjects
Brief Title: Safety, Tolerability, and Pharmacokinetics of Single Ascending Oral Doses of INV-101 in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inversago Pharma Inc. (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INV101-CL-101
Record Dates: First submitted 2020-08-24; First posted 2020-08-28 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pharmacokinetic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Fully blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Subjects will be randomized to receive either placebo or 20 mg INV-101
  Interventions: Drug: INV-101; Drug: Placebo
- Cohort 2 (Experimental): Subjects will be randomized to receive either placebo or 80 mg INV-101
  Interventions: Drug: INV-101; Drug: Placebo
- Cohort 3 (Experimental): Subjects will be randomized to receive either placebo or 160 mg INV-101
  Interventions: Drug: INV-101; Drug: Placebo
- Cohort 4 (Experimental): Subjects will be randomized to receive either placebo or 320 mg INV-101
  Interventions: Drug: INV-101; Drug: Placebo
- Cohort 5 (Experimental): Subjects will be randomized to receive either placebo or 500 mg INV-101
  Interventions: Drug: INV-101; Drug: Placebo

INTERVENTIONS:
Drug: INV-101 — Subjects will be randomized to receive INV-101 tablets
Drug: Placebo — Subjects will be randomized to receive placebo tablets

SUMMARY:
Single center, randomized, double-blinded, placebo-controlled, single ascending-dose study for the evaluation of the safety, tolerability, and PK following single oral doses of INV-101.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female
* Body mass index (BMI) within 18.5 kg/m2 to 30.0 kg/m2, inclusively; and body weight ≥60 kg
* Non- or ex-smoker
* Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination (including vital signs) and/or ECG, as determined by an investigator

Exclusion Criteria:

* Female who is pregnant or lactating
* Presence or history of significant gastrointestinal, liver or kidney disease, or surgery that may affect drug bioavailability
* History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
* Presence of clinically significant ECG abnormalities at the screening visit, as defined by medical judgment (maximum QTc of 450 for males and 470 for females)

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-01-16 (Actual); Study Completion 2021-05-16 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters - Maximum Concentration (Cmax) | 72 hours
  Cmax following single dose
Pharmacokinetic parameters - AUC | 72 hours
  AUC following single dose
Pharmacokinetic parameters - Half-live | 72 hours
  Half-live following single dose

SECONDARY OUTCOMES:
Adverse events | 72 hours
  Safety of INV-101 following single dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Altasciences, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No